CLINICAL TRIAL: NCT05501223
Title: Physician-initiated Medication Review in a Type 2 Diabetes Outpatient Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Karl Sebastian Johansson, Dr., PhD student, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P-2020-1012
Record Dates: First submitted 2021-08-03; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Polypharmacy
Keywords: Polypharmacy
MeSH Terms: interventions — Medication Review; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Standard care + medication review
  Interventions: Other: Medication review; Other: Standard care
- Control (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Medication review — 30-60 minutes extra consultation regarding the patients drugs
  Arms: Intervention
Other: Standard care — Standard care i.e. visit at the Dept. of Endocrinology.

SUMMARY:
Aiming to reduce polypharmacy in patients with type 2 diabetes by using physician-initiated medication reviews.

DETAILED DESCRIPTION:
Patients will be randomised to either standard care(annual visit at outpatient clinic) or standard care plus an intervention. The intervention is a medication consultation of 30-60 minutes that consist of a medication review and increased cross-sectoral communication. Follow-up is 6 months. Primary outcome are number of medications used, secondary outcomes are health related quality of life and persistance of medication changes.

ELIGIBILITY:
Inclusion Criteria:

1. DM2
2. 12 medications in the central prescription list

Exclusion Criteria:

1. inability to give written consent (e.g., inability to understand the intervention or language barriers);
2. active cancer or palliative treatment;
3. admitted to the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Number of medications used at baseline compared to number of medications used at follow-up. Resulting in a rate of medications used at baseline compared to follow-up i.e. no. medication at follow-up/no. at baseline. | 6 months
  The no. of medications used at baseline will be compared to the no. of medications used at follow-up. This will result in a rate i.e. no. at follow-up/no. at baseline which can be compared between groups resulting in a rate ratio. Medication usage is determined by number of medications listed in the central prescription list.

SECONDARY OUTCOMES:
EQ5D index score. (a Euro Quality of Life 5-dimension 5-level (EQ-5D-5L) scale). The score is retrieved by using the validated EQ5D questionnaire which translates to a corresponding EQ5D index score using country specific value sets. | 6 months
  Health related quality of life measured by EQ5D index score using Danish value sets (ranging from -0.7 (worst quality of life) to 1 (best quality of life)).

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark